CLINICAL TRIAL: NCT06455735
Title: 68Ga-JH04 PET/CT in Patients With Various Types of Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-JH04 PET/CT
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-04

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-JH04 PET/ CT (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-JH04. Tracer doses of 68Ga-JH04 will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-JH04
- 68Ga-FAPI/18F-FDG PET/ CT (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg 18F-FDG. Tracer doses of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-FAPI/18F-FDG

INTERVENTIONS:
Drug: 68Ga-JH04 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-JH04. Tracer doses of 68Ga-JH04 will be used to detect tumors by PET/CT.
  Arms: 68Ga-JH04 PET/ CT
Drug: 68Ga-FAPI/18F-FDG — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg 18F-FDG. Tracer doses of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Arms: 68Ga-FAPI/18F-FDG PET/ CT

SUMMARY:
As a novel radiotracer targeting fibroblast activation protein (FAP), 68Ga-JH04 is promising as an excellent imaging agent for various cancers. In this study, we observed the diagnostic performance of 68Ga-JH04 PET/CT in patients with different types of cancer, and compared its imaging results with those of 68Ga-FAPI or 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Carcinoma-associated fibroblasts (CAFs) are an integral part of the tumor microenvironment, and fibroblast activation protein (FAP), as a specific marker of CAFs, is overexpressed in more than 90% of epithelial malignant tumors' CAFs, with limited expression in normal tissues, making it an appropriate target for various tumors. Currently, several tracers targeting FAP for diagnostic purposes have been developed, such as 68Ga-FAPI-04, 68Ga-FAPI-02, showing high efficacy in tumor staging and restaging. As an emerging molecule targeting FAP, 68Ga-JH04, in this study, the diagnostic performance of 68Ga-JH04 PET/CT in patients with different types of cancer were observed. Its imaging results were compared with those of 68Ga-FAPI or 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

Various solid tumors with available histopathological findings Signed informed consent

Exclusion Criteria:

pregnant or lactational women who suffered from severe hepatic and renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-JH04 in Patients With Various Types of Cancer and comrared it with 68Ga-FAPI/18F-FDG PET/CT.

SECONDARY OUTCOMES:
SUV of tumors | through study completion, an average of 3 months
  Compare the SUV of tumors between 68Ga-JH04 PET/CT and 68Ga-FAPI/18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — The First Affiliated Hospital, Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No